CLINICAL TRIAL: NCT06180408
Title: Foot Spine Syndrome "RAFFET Syndrome" New Critical Implication in Clinical Biomechanics
Brief Title: Foot Spine Syndrome "RAFFET Syndrome"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Noha Khaled Shoukry (Other)
Responsible Party: Sponsor-Investigator, Noha Khaled Shoukry, lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Cairounivers
Record Dates: First submitted 2023-12-05; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Chronic Low-back Pain; Hallux Rigidus
MeSH Terms: conditions — Hallux Rigidus | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual therapy for the big toe (Experimental): Maitland mobilization (Grade 3,4), Mulligan mobilization with movement techniques, muscle energy techniques, manual therapy for plantar fascia, strengthening exercises and self-stretching exercises was performed
  Interventions: Other: manual therapy and exercise for the big toe
- lumbar stabilization exercise (Experimental): core training and myofascial release therapy
  Interventions: Other: lumbar stabilization exercise

INTERVENTIONS:
Other: manual therapy and exercise for the big toe — Maitland mobilization (Grade 3,4), Mulligan mobilization with movement techniques, muscle energy techniques, manual therapy for plantar fascia, strengthening exercises and self-stretching exercises was performed
  Arms: manual therapy for the big toe
Other: lumbar stabilization exercise — core training and myofascial release therapy
  Arms: lumbar stabilization exercise

SUMMARY:
case series aimed to describe a new clinical condition for the first time in the medical literature called Foot Spine Syndrome or "RAFFET Syndrome". This syndrome was reported in 11 patients (6 males and 5 females) out of 4000 patients with a history of chronic low back pain (CLBP) throughout 2 to 6 years in an outpatient clinic in Egypt from 2016 to 2022.

DETAILED DESCRIPTION:
Foot pain is usually derived from systemic disorder or local physical issues, such as tendonitis, arthritis, or bursitis. However, in some cases, pain in your foot may be linked to problems in your spine. This case series aimed to describe a new clinical condition for the first time in the medical literature called Foot Spine Syndrome or "RAFFET Syndrome". This syndrome was reported in 11 patients (6 males and 5 females) out of 4000 patients with a history of chronic low back pain (CLBP) throughout 2 to 6 years in an outpatient clinic in Egypt from 2016 to 2022. The patients suffered from CLBP that did not respond to physical therapy or any medication for long. They all had clinical spinal instability, hallux rigidus, foot abnormalities and tightness of hip flexors and adductors accompanied with weakness of hip extensors and abductors on the affected side. Manual therapy for the big toe including; Maitland mobilization (Grade 3,4), Mulligan mobilization with movement techniques, muscle energy techniques, manual therapy for plantar fascia, strengthening exercises and self-stretching exercises was performed.

ELIGIBILITY:
Inclusion Criteria:

* patients with a history of chronic low back pain (CLBP) did not respond to physical therapy or any medication for long. They all had clinical spinal instability, hallux rigidus, foot abnormalities and tightness of hip flexors and adductors accompanied with weakness of hip extensors and abductors on the affected side

Exclusion Criteria:

* any structural deformity (wedge fracture) or previous spinal surgeries. Spinal tumors or fracture or presence of active infection in the lumbar spine. Systematic disorder (Rheumatoid) Cauda equine lesion, the presence of any comorbidities such as hypertension, DM, hyperlipidemia, obesity, and any autoimmune disease, history of patients who suffered from cancer, unexplained weight loss, immunosuppression, prolonged use of steroids, intravenous drug use, urinary tract infection, pain that is increased or unrelieved by rest, fever, significant trauma related to age, bladder or bowel incontinence, urinary retention (with overflow incontinence), saddle anesthesia, loss of anal sphincter tone, major motor weakness in lower extremities, fever, and vertebral tenderness.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
numerical pain rating scale | three months
  considered the gold standard for back pain assessment
Oswestry disability index | three months
  It is a valid, reliable and responsive clinical tool used to determine the level of functional disability associated with CLBP

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No